CLINICAL TRIAL: NCT04743193
Title: Comparison of the Consumption of Sevoflurane in Two Different Concentrations and Two Different Currents During the Initial Period of Anesthesia in Patients Undergoing General Anesthesia With Minimal Flow
Brief Title: Different Low-flow Sevoflurane Anesthesia Techniques
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tahsin Şimşek, principal investigator, Kocaeli Derince Education and Research Hospital
Other Study IDs: 2020-514-169-13
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia
Keywords: inhalation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sevoflurane 8 %: In the initial phase, after reaching 1 (MAK) level with 1lt / min fresh gas flow and 8% sevoflurane concentration, anesthesia maintenance will be continued with 0.5 lt / min fresh gas flow and 2 -4% sevoflurane concentration with the target of 1 MAC.
  Interventions: Other: 8% sevoflurane low flow anesthesia
- sevoflurane 2.5 %: In the initial phase, after reaching 1 MAK level with 4 lt / min fresh gas flow and 2.5% sevoflurane concentration, anesthesia maintenance will be continued with 0.5 lt / min fresh gas flow and 2 -4% sevoflurane concentration with the target of 1 MAC.
  Interventions: Other: 2.5 %sevoflurane

INTERVENTIONS:
Other: 2.5 %sevoflurane — for 35 patients after reaching 1 MAK level with 4 lt / min fresh gas flow and 2,5% sevoflurane concentration in the initial phase, maintenance of anesthesia will be continued with 0.5 lt / min fresh gas flow and 2 -4% sevoflurane concentration with the target of 1 minimum alveolar concentration
  Groups: sevoflurane 2.5 %
Other: 8% sevoflurane low flow anesthesia — For 35 patients after reaching 1 (MAC) level with 1 lt / min fresh gas flow and 8% sevoflurane concentration in the initial phase, maintenance of anesthesia will be continued with 0.5 lt / min fresh gas flow and 2 -4% sevoflurane concentration, targeting 1 MAC. .
  Groups: sevoflurane 8 %

SUMMARY:
After reaching 1 MAC level with 4 lt / min fresh gas flow and 2.5% sevoflurane concentration in the initial stage in 35 patients, anesthesia maintenance will be continued with 0.5 lt / min fresh gas flow and 2 -4% sevoflurane concentration with the target of 1 MAC. For 35 patients, after reaching 1 (MAC) level with 1 lt / min fresh gas flow and 8% sevoflurane concentration in the initial phase, maintenance of anesthesia will be continued with 0.5 lt / min fresh gas flow and 2 -4% sevoflurane concentration, targeting 1 MAC.

DETAILED DESCRIPTION:
The primary aim of this study is to compare the instantaneous and total consumption of sevoflurane using 2 different concentrations and different minute / fresh gas flow to fill the system in the initial phase of anesthesia. Its secondary purpose is to compare the depth of anesthesia and hemodynamic parameters between the two groups.

A total of 70 patients between the ages of 18-65 will be included in the study.in 2.5 % sevoflurane grup After reaching 1 MAC level with 4 lt / min fresh gas flow and 2.5% sevoflurane concentration in the initial stage in 35 patients, anesthesia maintenance will be continued with 0.5 lt / min fresh gas flow and 2 -4% sevoflurane concentration with the target of 1 MAC. in sevoflurane 8 % group for 35 patients, after reaching 1 (MAC) level with 1 lt / min fresh gas flow and 8% sevoflurane concentration in the initial phase, maintenance of anesthesia will be continued with 0.5 lt / min fresh gas flow and 2 -4% sevoflurane concentration with the target of 1 MAC. . The depth of anesthesia for both groups will be measured by the Bispectral Index (BIS). BIS values between 40 and 60 are appropriate values for general anesthesia, for this value 1 MAC sevoflurane inhalation anesthesia and remifentanil infusion (0.1-0.3mcg / kg / min) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65
* ASA1,2,3 group patients
* Patients under general anesthesia
* Patients scheduled for elective surgery

Exclusion Criteria:

* The patient's refusal to participate in the study
* Patients with less than 90 minutes of total anesthesia time
* Patients whose total anesthesia time exceeds 180 minutes

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Patients between the ages of 18-65
  * ASA1,2,3 group patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
sevoflurane versus desflurane | the study will comlete in one month
  To compare the instant and total consumption of sevoflurane using 2 different concentrations and different minute / fresh gas flow to fill the system in the initial phase of anesthesia.

SECONDARY OUTCOMES:
sevoflurane | studdy will complete in one month
  Its secondary purpose is to compare the depth of anesthesia and hemodynamic parameters between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Tahsin Şimşek, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided